CLINICAL TRIAL: NCT01802008
Title: Comparison of Adenoma Detection and Miss Rates at Colonoscopy Associated With a Six-minute Withdrawal Time vs a Three-minute Withdrawal Time
Brief Title: Comparison of Adenoma Detection Miss Rates at Colonoscopy Associated With Different Withdrawal Times
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Subhas Banerjee, Principle Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-25203
Record Dates: First submitted 2013-02-27; First posted 2013-03-01 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Adenoma and/or Adenocarcinoma; Adenoma
Keywords: Polyp/adenoma detection rate; Polyp/adenoma miss rate; Colonoscopy withdrawal time
MeSH Terms: conditions — Adenoma; Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 3-minute withdrawal time (Active Comparator): For subjects randomized to the 3-minute withdrawal time, advancement to the cecum will be followed by segmental withdrawal in each of 3 segments of the examined colon. Each segment will be examined over 1 minute, followed by a "second look" over each segment over 2 minutes by the same endoscopist.
  Interventions: Procedure: 3-minute withdrawal time
- 6-minute withdrawal time (Active Comparator): For subjects randomized to the 6-minute withdrawal, advancement to the cecum will be followed by segmental withdrawal in each of 3 segments of the examined colon. Each segment will be examined over 2 minutes, followed by a "second look" over each segment over 2 minutes by the same endoscopist.
  Interventions: Procedure: 6-minute withdrawal time

INTERVENTIONS:
Procedure: 3-minute withdrawal time — For subjects randomized to the 3-minute withdrawal time, advancement to the cecum will be followed by segmental withdrawal in each of 3 segments of the examined colon. Each segment will be examined over 1 minute, followed by a "second look" over each segment over 2 minutes by the same endoscopist.
  Arms: 3-minute withdrawal time
Procedure: 6-minute withdrawal time — For subjects randomized to the 6-minute withdrawal, advancement to the cecum will be followed by segmental withdrawal in each of 3 segments of the examined colon. Each segment will be examined over 2 minutes, followed by a "second look" over each segment over 2 minutes by the same endoscopist.
  Arms: 6-minute withdrawal time

SUMMARY:
The objective of this study is to determine the optimal withdrawal time for colonoscopy. A 6-minute withdrawal time is currently the standard of care but has only been evaluated in an observational fashion. The investigators believe that this should be validated in a standardized fashion. If the benefits of a 6 minute withdrawal are proven in this study (ie a low polyp/adenoma miss rate and a high polyp/adenoma detection rate), then this will support widespread adoption of a 6 minute withdrawal as the standard of care. This in turn may decrease the occurence of 'interval colon cancers', which are early colon cancers arising in subjects despite their having undergone colonoscopy. Our hypothesis is that the polyp/adenoma detection rate will be unacceptably low and the polyp/adenoma miss rate will be unacceptably high in the 3-minute withdrawal group when compared to the 6-minute withdrawal group.

DETAILED DESCRIPTION:
Eligible patients will be randomized to colonoscopy with either a 6-minute withdrawal time or a 3-minute withdrawal time. Patients will then undergo colonoscopy. All colonoscopies will be performed by a GI attending (standard of care). The colonoscopy is typically performed under conscious sedation using medications such as fentanyl and midazolam for comfort (standard of care). Occasional patients undergo colonoscopy under general anesthesia. For all patients, advancement of the colonoscope to the cecum will be followed by segmental withdrawal of the colonoscope in each of 3 segments of the examined colon (right side of colon, transverse colon and left side of colon). Following examination of each individual segment, the colonoscope will be readvanced to the proximal end of the segment and a 2 minute withdrawal will be re-performed. For those randomized to the 6-minute withdrawal each segment will be examined over 2 minutes, followed by a "second look" over each segment over 2 minutes by the same endoscopist. For those randomized to the 3-minute withdrawal time, advancement to the cecum will also be followed by segmental withdrawal in each of 3 segments of the examined colon. Each segment will be examined over 1 minute, followed by a "second look" over each segment over 2 minutes by the same endoscopist. All patients will therefore undergo a second look colonoscopy with a 6-minute withdrawal time ('de-facto' standard of care). Polyp/adenoma detection and miss rates will then be calculated and compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Already scheduled for colonoscopy

Exclusion Criteria:

* Age < 18
* Pregnant women
* Mentally disabled
* Decisionally challenged
* Cancer subjects
* Healthy volunteers
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Polyp/Adenoma Detection Rate | This will be calculated up to one week after data collection.
  Polyp/adenoma detection rate will be calculated for each segment of the tandem colonoscopy- this will be calculated as the number of polyps/adenomas that are discovered and resected for each segment of the tandem colonoscopy.
Polyp/adenoma Miss Rate | Polyp/adenoma miss rate will be calculated up to one week after data collection.
  Polyp/adenoma miss rate will be calculated for each segment of the tandem colonoscopy- this will be calculated as the number of polyps/adenomas that are discovered and resected on the tandem portion of each segment of the colonoscopy, divided by the total number of polyps/adenomas that are discovered/resected.

CONTACTS AND LOCATIONS:
Overall Officials: Subhas Banerjee, M.D., Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Veterans Administration Hospital (Palo Alto), Palo Alto, California
  - Stanford University, Palo Alto, California

REFERENCES:
- [Derived] Kumar S, Thosani N, Ladabaum U, Friedland S, Chen AM, Kochar R, Banerjee S. Adenoma miss rates associated with a 3-minute versus 6-minute colonoscopy withdrawal time: a prospective, randomized trial. Gastrointest Endosc. 2017 Jun;85(6):1273-1280. doi: 10.1016/j.gie.2016.11.030. Epub 2016 Dec 6. PMID 27931951